CLINICAL TRIAL: NCT06428669
Title: The Effect of Nitropaste in Chest Masculinizing Surgery: Randomized, Prospective Trial
Brief Title: Effect of Nitropaste in Chest Masculinizing Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, John Stranix, Assistant Professor, Department of Plastic Surgery, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSR220217
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Gender Dysphoria
Keywords: Gender affirming surgery; Chest masculinizing Surgery; Nitropaste; Wound healing
MeSH Terms: conditions — Gender Dysphoria | interventions — Nitroglycerin; Ointments

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- No nitropaste group (No Intervention): Participants get standard of care chest masculinizing surgery utilizing double incision and free nipple grafting surgery. They will get standard dressing applied, which includes Xeroform bolster over the nipple grafts + Tegederm over the bolster and surgical site and instructed not to remove the dressing until they come to clinic on POD5 for bolster take down.
- Nitropaste group (Experimental): Participants get standard of care chest masculinizing surgery utilizing double incision and free nipple grafting surgery. They will then get 2 packets of nitropaste applied (1 on each chest) around the free nipple graft and surgical sites. They will then get standard dressing applied, which includes Xeroform bolster over the nipple grafts + Tegederm over the bolster and surgical site and instructed not to remove the dressing until they come to clinic on POD5 for bolster take down.
  Interventions: Drug: Nitro-Bid 2 % Topical Ointment

INTERVENTIONS:
Drug: Nitro-Bid 2 % Topical Ointment — Intervention group will get 30mg of Nitro-Bid topical ointment applied over the chest (15mg/ 1 packet on each side) one time intra-operatively
  Arms: Nitropaste group

SUMMARY:
Nitropaste is a topical agent that contains 2% nitroglycerin. It is an effective vascular smooth dilator, with more powerful effect on venous vasculature than arterial vasculature. While its main indication is for angina pectoris, there have been many studies showing improved survival of axial and random pattern flaps. Furthermore, recent clinical studies highlight significantly decreased mastectomy flap wound complication and need for sharp debridement. Nitropaste has low rates of side effects and is very well tolerated in general. To this date, there's no study that investigates its utility on patients who are undergoing chest masculinizing surgery. The purpose of this study is to investigate the potential utility of nitropaste in reducing rates of wound complications in patients undergoing chest masculinizing surgery.

DETAILED DESCRIPTION:
Nitropaste is a topical agent that contains 2% nitroglycerin. It is an effective vascular smooth dilator, with more powerful effect on venous vasculature than arterial vasculature. While its main indication is for angina pectoris, there have been many studies showing improved survival of axial and random pattern flaps. Furthermore, recent clinical studies highlight significantly decreased mastectomy flap wound complication and need for sharp debridement. Nitropaste has low rates of side effects and is very well tolerated in general. To this date, there's no study that investigates its utility on patients who are undergoing chest masculinizing surgery. The purpose of this study is to investigate the potential utility of nitropaste in reducing rates of wound complications in patients undergoing chest masculinizing surgery utilizing double incision with free nipple grafting technique. The investigators will conduct a prospective, randomized, single-blinded study and compare nitropaste vs. no nitropaste on mastectomy flaps. Nitropaste will be applied intraoperatively and the patients will not have to re-apply it. Follow up will occur on post-op day 5, 2 weeks, and 6 weeks during their routine postop visits. A study coordinator will document the condition of free nipple grafts and any other wounds at surgical site if present, which will be the primary outcome. Any complications including hematoma, seroma, infection, hypertrophic scarring, need for sharp debridement, 30 day ED visit or admission rates will be documented as secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Any adult (18 or older) patients of any gender identity who are undergoing chest masculinizing surgery with double incision and free nipple grafting.

Exclusion Criteria:

* Minor patients (younger than 18)
* Anyone who's not getting free nipple grafting
* Anyone who's not utilizing double incision pattern
* Prisoners, anyone who is allergic to nitropaste
* Anyone who is taking phosphodiesterase inhibitor (ex)Sildenafil, tadalafil, vardenafil)
* Anyone who's taking soluble guanylate cyclase stimulator riociguatdz

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Free Nipple Graft Take | Will be assessed at 5 days, 2 weeks, 6 weeks post-op
  Rate of partial nipple graft loss (0-50%, 50% or more) or Complete nipple graft loss
Wounds | Will be assessed at 5 days, 2 weeks, 6 weeks post-op
  Rate of superficial wound, deep wound, delayed wound healing

SECONDARY OUTCOMES:
Complications | Will be tracked up until 3 months post-op
  hematoma, seroma, infection, hypertrophic scarring
Sharp debridement | Will be tracked up until 3 months post-op
  Need for any sharp debridement (office or OR)
Revision | Will be tracked up until 3 months post-op
  Need for any revision
Readmission | Will be tracked 30 days
  30 day ED or inpatient admission rate

CONTACTS AND LOCATIONS:
Overall Officials: John T Stranix, MD, Principal Investigator — UVA
Locations (1):
- University of Virginia Medical Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park RH, Pawly J, Grogan G, DeVito RG, Ke BG, Behar BJ, Stranix JT. Topical Nitropaste Reduces Partial Free Nipple Graft Loss in Gender Affirming Mastectomy: A Randomized Controlled Trial. Plast Reconstr Surg. 2026 Feb 2. doi: 10.1097/PRS.0000000000012874. Online ahead of print. PMID 41628614

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT06428669/Prot_SAP_000.pdf